CLINICAL TRIAL: NCT05736042
Title: Microinterventional Endocapsular Nuclear Fragmentation Assisted Cataract Surgery Versus Conventional Phacoemulsification Using Divide-and-conquer: a Randomized Controlled Trial
Brief Title: Microinterventional Endocapsular Nuclear Fragmentation Assisted Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oogziekenhuis Rotterdam (Other)
Collaborators: Stichting Wetenschappelijk Onderzoek Het Oogziekenhuis Prof.dr H.J. Flieringa (Unknown); Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OZR-2022-07; NL83139.078.22 (Other: CCMO)
Record Dates: First submitted 2023-01-31; First posted 2023-02-21 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Nuclear Cataract
Keywords: LOCS III grade 5 or more

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lens fragmentation with miLOOP (Experimental): Phacoemulsification with adjunctive lens fragmentation with the microinterventional microfilament loop device (miLOOP)
  Interventions: Device: Lens fragmentation
- Controls (No Intervention): Phacoemulsification alone (no adjunctive lens fragmentation)

INTERVENTIONS:
Device: Lens fragmentation — Lens fragmentation with the microinterventional microfilament loop device (miLOOP)
  Arms: Lens fragmentation with miLOOP

SUMMARY:
Rationale: In cataract surgery, fragmentation of a hard nucleus requires relatively much ultrasound energy. It is suspected that the level of energy used is associated with the degree of corneal endothelial loss. Recently, it was demonstrated that with miLOOP (Zeiss Meditec) assisted nuclear fragmentation ultrasound energy can be substantially reduced.

Objective: To compare miLOOP assisted cataract surgery and conventional surgery with respect to the energy needed for phacoemulsification and loss of corneal endothelial cells.

Study design: Randomized, controlled trial. Study population: Patients with nuclear cataract of a grade ≥ 5. Intervention: Microinterventional endocapsular nuclear fragmentation. Main study parameters: Cumulative dispersed ultrasound energy (CDE) and endothelial cell loss.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Informed consent.
* Advanced visually significant nuclear sclerosis grade ≥ 5 (LOCS III).

Exclusion Criteria:

* Endothelial cell density (ECD) < 1500 mm-2.
* Corneal opacification (any cause).
* Corneal surgery or trauma.
* Implant lens.
* Refraction surgery.
* Prior glaucoma surgery.
* Pseudoexfoliation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Ultrasound cumulative dispersed energy (CDE) | During surgery
  Phaco energy (Centurion, Alcon)
Change of corneal endothelial cell density (ECD) | Preoperative and at 3 months
  Central cell density will be assessed

SECONDARY OUTCOMES:
Procedure time | During surgery
  Total sugery time
Peri-operative complications | During surgery
  Any complications during surgery
Postoperative complications | Up to 3 months
  Any complications after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Oogziekenhuis Rotterdam, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No